CLINICAL TRIAL: NCT01239173
Title: Reliving the Traumatic Event in Posttraumatic Stress Disorder: An Emotional Memory Reactivation Pathology? An fMRI Study
Brief Title: Emotional Memory Reactivation in Posttraumatic Stress Disorder
Acronym: VIVITRAU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped by promoter for lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOM06075/ P060226
Record Dates: First submitted 2010-10-25; First posted 2010-11-11 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic stress disorder; functional Magnetic Resonance Imaging; Amygdala; emotion regulation; memory
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Emotional Regulation | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Post-traumatic stress disorder patient receiving propanolol 90 min before the emotional memory reactivation and the anatomical and functional exploration in fMRI
  Interventions: Drug: AVLOCARDYL
- 2 (Placebo Comparator): Post-traumatic stress disorder receiving placebo 90 min before the emotional memory reactivation and the anatomical and functional exploration in fMRI
  Interventions: Drug: Placebo
- 3 (Active Comparator): Controls receiving propanolol 90 min before the emotional memory reactivation and the anatomical and functional exploration in fMRI
  Interventions: Drug: AVLOCARDYL
- 4 (Placebo Comparator): Controls receiving placebo 90 min before the emotional memory reactivation and the anatomical and functional exploration in fMRI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVLOCARDYL — A grip of 2 tablets of 20 mg each took 90 min before the emotional memory reactivation and the anatomical and functional exploration in fMRI
  Arms: 1
Drug: Placebo — A grip of 2 tablets of 20 mg each took 90 min before the emotional memory reactivation and the anatomical and functional exploration in fMRI
  Arms: 2
Drug: AVLOCARDYL — A grip of 2 tablets of 20 mg each took 90 min before the emotional memory reactivation and the anatomical and functional exploration in fMRI
  Arms: 3
Drug: Placebo — A grip of 2 tablets of 20 mg each took 90 min before the emotional memory reactivation and the anatomical and functional exploration in fMRI
  Arms: 4

SUMMARY:
Converging lines of evidence have implicated the amygdala in the pathophysiology of posttraumatic stress disorder.

The primary purpose of our study is to assess the effect of propanolol, a beta adrenergic antagonism, on amygdala activation during a symptom provocation state in traumatized subjects with and without posttraumatic stress disorder.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a type of anxiety disorder that's triggered by an extremely traumatic event. Traumatic events that may trigger PTSD include violent personal assaults, accidents, natural or human-caused disasters, or military combat. Converging lines of evidence have implicated the amygdala in the pathophysiology of posttraumatic stress disorder.

Initially based on animal studies, the idea that memory for emotional material in humans is modulated by the noradrenergic system and by the amygdala, has received a strong support over the last decade. Evidence mainly comes from studies investigating the effect of emotion on encoding processes (Mc GAUGH, 2000). In that view, propranolol has been used somewhat successfully shortly after trauma to reduce the development of PTSD symptoms (Pitman et al., 2002; VAIVA et al., 2003). As already mentioned, "reconsolidation" studies developed in rats provide treatment strategies that can be used long after PTSD induction. Recent evidence indicates that consolidated long-term memory in human can also be influenced by events delivered after memory reactivation (Walker et al., 2003; HUPBACH et al., 2007), suggesting that human memory can be retroactively altered by treatments delivered in conjunction with memory reactivation. This seems to be confirmed by an as yet unpublished human based study that suggests that propranolol may impair reconsolidation of conditioned fear-response (Miller et al., 2004) The primary purpose of our study is to assess the effect of propanolol, a beta adrenergic antagonism, on amygdala activation during a symptom provocation state in traumatized subjects with and without posttraumatic stress disorder. One Functional magnetic resonance imaging (fMRI) will be performed (week 1) in 32 patients with PTSD and 32 controls (exposure to a traumatic event without PTSD) to examine amygdala activation during a provocation state.

One half of the patients with PTSD and one half of the controls will receive propranolol prior the fMRI under double blind condition.

In addition, a cognitive test battery will be performed (screening, week 0, 1, 2) before the fRMI acquisition and at follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients of French mother language
* Right-handed patients
* Signature of the consent

Patients:

* Patients whose diagnosis of PTSD according to the criteria of the DSM IV-TR is established
* PTSD whose evolution is not chronic
* Established PTSD : Symptoms presents for at least 1 month
* PTSD consecutive to a unique traumatic event

Controls :

* The healthy controls will have sudden a traumatism of the same nature or the nature comparable to that of the patients suffering from PTSD, but they will not have developed pathology
* Subjects having undergone a traumatism dating less than 3 months
* Examples of traumatic events: aggression, accident of the public highway, the occupational accident

Exclusion Criteria:

* The PTSD consecutive to several traumatic events
* Patients treated by a substance crossing the blood-brain barrier (with the exception of the antidepressants of the family of the ISRS which can be indicated in the treatment of PTSD)
* Histories of epilepsy or significant loss of consciousness of any origin, including post-traumatic
* Any psychiatric or somatic significant pathology
* The psychiatric histories in particular of suicide attempt
* The pregnant or breast-feeding women
* Contraindications in the propanolol
* Consumption of psychoactive drugs detected in urines
* Excessive alcohol consumption
* The persons not being capable of understanding or of reading the information describing the study
* The patients refusing to sign the form of consent of participation for the study
* The left-handed or ambidextrous patients
* The patients without the general regime of the health insurance
* The patients under guardianship or incapable major
* The patients who will not be capable of supplying a documentary evidence of identity the day of the inclusion
* Contraindication in the practice of a MRI
* The patients or the controls refusing the medical and psychiatric balance assessment of screening cannot participate in the study
* Strong probability of not compliance to the protocol or of abandonment in the course of study
* Taking of a speechless medicine, in particular beta-blocking
* Participating in phase of exclusion from a previous study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Effect of propanolol, a beta adrenergic antagonism, on amygdala activation during a symptom provocation state in traumatized subjects with and without posttraumatic stress disorder | 34 days

SECONDARY OUTCOMES:
Comparison of propranolol therapeutic effects versus placebo on symptom provocation state in traumatized subjects with and without posttraumatic stress disorder | 34 days
Comparison of activated neuronal networks when a patient remember a pleasant , unpleasant or traumatic event | 34 days
Comparison of emotional status of traumatized subjects with and without posttraumatic stress disorder | 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Siegfried Peretti, MD, PhD, Principal Investigator — Saint-Antoine hospital, Psychiatry unit, ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS
Locations (1):
- Saint-Antoine Hospital, Psychiatriy unit, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Adler SA, Wilk A, Rovee-Collier C. Reinstatement versus reactivation effects on active memory in infants. J Exp Child Psychol. 2000 Feb;75(2):93-115. doi: 10.1006/jecp.1999.2531. PMID 10620375
- [Background] Blanchard EB, Hickling EJ, Taylor AE, Forneris CA, Loos W, Jaccard J. Effects of varying scoring rules of the Clinician-Administered PTSD Scale (CAPS) for the diagnosis of post-traumatic stress disorder in motor vehicle accident victims. Behav Res Ther. 1995 May;33(4):471-5. doi: 10.1016/0005-7967(94)00064-q. PMID 7755537
- [Background] Botreau F, El Massioui N, Cheruel F, Gisquet-Verrier P. Effects of medial prefrontal cortex and dorsal striatum lesions on retrieval processes in rats. Neuroscience. 2004;129(3):539-53. doi: 10.1016/j.neuroscience.2004.08.032. PMID 15541876
- [Background] Boujabit M, Bontempi B, Destrade C, Gisquet-Verrier P. Exposure to a retrieval cue in rats induces changes in regional brain glucose metabolism in the amygdala and other related brain structures. Neurobiol Learn Mem. 2003 Jan;79(1):57-71. doi: 10.1016/s1074-7427(02)00010-2. PMID 12482680
- [Background] Brunet A, Orr SP, Tremblay J, Robertson K, Nader K, Pitman RK. Effect of post-retrieval propranolol on psychophysiologic responding during subsequent script-driven traumatic imagery in post-traumatic stress disorder. J Psychiatr Res. 2008 May;42(6):503-6. doi: 10.1016/j.jpsychires.2007.05.006. Epub 2007 Jun 22. PMID 17588604
- [Background] Dirikx T, Hermans D, Vansteenwegen D, Baeyens F, Eelen P. Reinstatement of extinguished conditioned responses and negative stimulus valence as a pathway to return of fear in humans. Learn Mem. 2004 Sep-Oct;11(5):549-54. doi: 10.1101/lm.78004. PMID 15466307
- [Background] Ferry B, McGaugh JL. Clenbuterol administration into the basolateral amygdala post-training enhances retention in an inhibitory avoidance task. Neurobiol Learn Mem. 1999 Jul;72(1):8-12. doi: 10.1006/nlme.1998.3904. PMID 10371711
- [Background] Giles J. Beta-blockers tackle memories of horror. Nature. 2005 Jul 28;436(7050):448-9. doi: 10.1038/436448a. No abstract available. PMID 16049437
- [Background] Gisquet-Verrier P, Botreau F, Venero C, Sandi C. Exposure to retrieval cues improves retention performance and induces changes in ACTH and corticosterone release. Psychoneuroendocrinology. 2004 May;29(4):529-56. doi: 10.1016/s0306-4530(03)00085-4. PMID 14749097
- [Background] Herz RS. Are odors the best cues to memory? A cross-modal comparison of associative memory stimuli. Ann N Y Acad Sci. 1998 Nov 30;855:670-4. doi: 10.1111/j.1749-6632.1998.tb10643.x. PMID 9929669
- [Background] Maheu FS, Joober R, Beaulieu S, Lupien SJ. Differential effects of adrenergic and corticosteroid hormonal systems on human short- and long-term declarative memory for emotionally arousing material. Behav Neurosci. 2004 Apr;118(2):420-8. doi: 10.1037/0735-7044.118.2.420. PMID 15113269
- [Background] Przybyslawski J, Roullet P, Sara SJ. Attenuation of emotional and nonemotional memories after their reactivation: role of beta adrenergic receptors. J Neurosci. 1999 Aug 1;19(15):6623-8. doi: 10.1523/JNEUROSCI.19-15-06623.1999. PMID 10414990
- [Background] Quirarte GL, Roozendaal B, McGaugh JL. Glucocorticoid enhancement of memory storage involves noradrenergic activation in the basolateral amygdala. Proc Natl Acad Sci U S A. 1997 Dec 9;94(25):14048-53. doi: 10.1073/pnas.94.25.14048. PMID 9391150
- [Background] Sara SJ. Retrieval and reconsolidation: toward a neurobiology of remembering. Learn Mem. 2000 Mar-Apr;7(2):73-84. doi: 10.1101/lm.7.2.73. No abstract available. PMID 10753974
- [Background] Simson PE, Naylor JC, Gibson B, Schneider AM, Levin D. Dose-sensitive excitation and inhibition of spontaneous amygdala activity by propranolol. Pharmacol Biochem Behav. 2001 May-Jun;69(1-2):85-92. doi: 10.1016/s0091-3057(01)00503-2. PMID 11420072
- [Background] Strange BA, Dolan RJ. Beta-adrenergic modulation of emotional memory-evoked human amygdala and hippocampal responses. Proc Natl Acad Sci U S A. 2004 Aug 3;101(31):11454-8. doi: 10.1073/pnas.0404282101. Epub 2004 Jul 21. PMID 15269349
- [Background] Taylor F, Cahill L. Propranolol for reemergent posttraumatic stress disorder following an event of retraumatization: a case study. J Trauma Stress. 2002 Oct;15(5):433-7. doi: 10.1023/A:1020145610914. PMID 12392232
- [Background] Vaiva G, Ducrocq F, Jezequel K, Averland B, Lestavel P, Brunet A, Marmar CR. Immediate treatment with propranolol decreases posttraumatic stress disorder two months after trauma. Biol Psychiatry. 2003 Nov 1;54(9):947-9. doi: 10.1016/s0006-3223(03)00412-8. PMID 14573324
- [Background] van Stegeren AH, Everaerd W, Cahill L, McGaugh JL, Gooren LJ. Memory for emotional events: differential effects of centrally versus peripherally acting beta-blocking agents. Psychopharmacology (Berl). 1998 Aug;138(3-4):305-10. doi: 10.1007/s002130050675. PMID 9725752
- [Background] van Stegeren AH, Goekoop R, Everaerd W, Scheltens P, Barkhof F, Kuijer JP, Rombouts SA. Noradrenaline mediates amygdala activation in men and women during encoding of emotional material. Neuroimage. 2005 Feb 1;24(3):898-909. doi: 10.1016/j.neuroimage.2004.09.011. PMID 15652324